CLINICAL TRIAL: NCT02350959
Title: Evaluation of Adverse Plaque Characteristics in Coronary Computed Tomography Angiography Using Combined Near Infrared Spectroscopy With Intravascular Ultrasound [CITRUS Study]
Brief Title: Adverse Plaque Characteristics in CCTA and TVC Imaging
Acronym: CITRUS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Insurance Service Ilsan Hospital (Other)
Responsible Party: Principal Investigator, Sanghoon Shin, Director, Clinical Research, National Health Insurance Service Ilsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-11-022
Record Dates: First submitted 2015-01-16; First posted 2015-01-30 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Plaque
Keywords: Plaque; coronary computed tomography angiography
MeSH Terms: conditions — Plaque, Amyloid | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose statin (Experimental): In high dose statin group, atorvastatin 40mg will be used
  Interventions: Drug: Atorvastatin
- Moderate dose statin (Active Comparator): in moderate dose statin group, atorvastatin 10mg will be used
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — in moderate dosea statin group, atorvastatin 10mg will be used and maintained until follow up angiography
  Arms: Moderate dose statin
Drug: Atorvastatin — in high dose statin group, atorvastatin 40mg will be used and maintained until follow up angiography
  Arms: High dose statin

SUMMARY:
The present study is intended to assess the vulnerability of plaques seen on CCTA by means of TVC Imaging System and to make comparisons between plaques with adverse plaque characteristics and ones without adverse plaque characteristics in terms of plaque volume and lipid core contents.

DETAILED DESCRIPTION:
This study is to be conducted in two phases - Phases 1 and 2. In Phase 1, the vulnerability of plaques seen on CCTA will be assessed with TVC Imaging System, and the plaque volume and lipid core contents of plaques with versus without adverse plaque characteristics will be compared. For the purpose of this study, the study of this phase will be a cross-sectional study in which the shapes of vulnerable plaques seen on CCTA will be compared to their vulnerability visualized by the TVC Imaging System.

In Phase 2, the patients with multi-vessel (polyvascular) disease of those participating in Phase 1 will be included, and the study of this phase will be a longitudinal study in which serial TVC imaging will be performed for non-target vessels, and any differences in changes of plaque vulnerability when treated with moderate-dose versus high-dose statin will be comparatively analyzed. The purpose of the present study is to determine whether there are any significant differences in changes of plaque volume and stability when treated with high-dose versus moderate-dose statin.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 years of older
2. Patients with typical chest pain or evidences of myocardial ischemia (e.g., stable, unstable angina, silent ischemia and positive functional study or reversible changes in the electrocardiogram (ECG) consistent with ischemia
3. Patients with signed informed consent
4. Confirmed coronary artery disease in computed tomography

Exclusion Criteria:

1. The past history of coronary artery disease (e.g., myocardial infarction, percutaneous coronary intervention (PCI), coronary artery bypass graft surgery (CABG), etc.)
2. Less than 2-year life expectancy due to non-cardiac disease
3. If the subject cannot voluntarily agree in writing to participate in this study
4. If the subject is currently participating in any other study with another investigational drug or medical device
5. Allergic reaction to iodinated contrast media
6. Significant renal dysfunction (Serum creatinine > 1.5 mg/dl) 7 Heart rate ≥ 80 beats per minute even after treatment with a heart rate lowering medication which disable to take CCTA

8. Contraindications of either β blockers or nitroglycerin 9. The past history of complex congenital heart disease 10. Pregnant women or women with potential childbearing 11. Body mass index (BMI) exceeding 35 12. Irregular heartbeats which disable to take CCTA 13. Contraindications of statin due to hypersensitivity, past history of serious complication such as myopathy or increased liver enzyme more than 3 times of normal upper limit

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
the change of max LCBI(4mm): Lipid core burden index in 4 mm | 1 year
  The primary endpoint for this study is the change of max LCBI(4mm) between initial and follow up angiography in non-target vessel
Correlation between vulnerable plaque on CT and max LCBI(4mm) | maximum duration of 3 months between CT and NIRS
  The other primary endpoint of this study is Vessel level correlation of vulnerable plaque on CT and LCBI(4mm)

SECONDARY OUTCOMES:
the change of presence of maxLCBI(4mm) > 500 | 1 year
  vessel level comparison between initial and follow up angiography in non-target vessel
the change of CT plaque vulnerability | 2years
  the change of Positive remodeling, Low attenuation plaque, Spotty calcification

CONTACTS AND LOCATIONS:
Overall Officials: Sanghoon Shin, M.D., Principal Investigator — National Health Insurance Service Ilsan Hospital
Locations (1):
- National Health Insurance Service Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] de Boer SP, Brugaletta S, Garcia-Garcia HM, Simsek C, Heo JH, Lenzen MJ, Schultz C, Regar E, Zijlstra F, Boersma E, Serruys PW. Determinants of high cardiovascular risk in relation to plaque-composition of a non-culprit coronary segment visualized by near-infrared spectroscopy in patients undergoing percutaneous coronary intervention. Eur Heart J. 2014 Feb;35(5):282-9. doi: 10.1093/eurheartj/eht378. Epub 2013 Sep 12. PMID 24037276
- [Background] Yonetsu T, Suh W, Abtahian F, Kato K, Vergallo R, Kim SJ, Jia H, McNulty I, Lee H, Jang IK. Comparison of near-infrared spectroscopy and optical coherence tomography for detection of lipid. Catheter Cardiovasc Interv. 2014 Nov 1;84(5):710-7. doi: 10.1002/ccd.25084. Epub 2013 Jul 16. PMID 23785015
- [Background] Madder RD, Goldstein JA, Madden SP, Puri R, Wolski K, Hendricks M, Sum ST, Kini A, Sharma S, Rizik D, Brilakis ES, Shunk KA, Petersen J, Weisz G, Virmani R, Nicholls SJ, Maehara A, Mintz GS, Stone GW, Muller JE. Detection by near-infrared spectroscopy of large lipid core plaques at culprit sites in patients with acute ST-segment elevation myocardial infarction. JACC Cardiovasc Interv. 2013 Aug;6(8):838-46. doi: 10.1016/j.jcin.2013.04.012. Epub 2013 Jul 17. PMID 23871513
- [Background] Jaguszewski M, Klingenberg R, Landmesser U. Intracoronary Near-Infrared Spectroscopy (NIRS) Imaging for Detection of Lipid Content of Coronary Plaques: Current Experience and Future Perspectives. Curr Cardiovasc Imaging Rep. 2013;6(5):426-430. doi: 10.1007/s12410-013-9224-2. PMID 24098825
- [Background] Pu J, Mintz GS, Brilakis ES, Banerjee S, Abdel-Karim AR, Maini B, Biro S, Lee JB, Stone GW, Weisz G, Maehara A. In vivo characterization of coronary plaques: novel findings from comparing greyscale and virtual histology intravascular ultrasound and near-infrared spectroscopy. Eur Heart J. 2012 Feb;33(3):372-83. doi: 10.1093/eurheartj/ehr387. Epub 2011 Oct 20. PMID 22019821